CLINICAL TRIAL: NCT00669552
Title: Intracardiac T-wave Alternans and Ischemia During Percutaneous Coronary Interventions
Brief Title: Intracardiac T-wave Alternans and Ischemia
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jose M. Dizon, Assoc Professor of Clinical, Department of Medicine Cardiology, Columbia University
Other Study IDs: AAAC6715
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medtronic defibrillator: Patients undergoing a percutaneous coronary intervention (PCI) with an implanted Medtronic defibrillator with the capability of telemetry of the intracardiac signal.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI previously electively scheduled.

SUMMARY:
T-wave alternans is a test that looks at microvolt changes in the T-wave on a beat to beat basis. The presence or absence of such changes has been shown to predict or exclude future arrhythmic events. The mechanism of T-wave alternans is unclear, but may relate to calcium metabolism in the heart, and may be affected by conditions such as ischemia or heart failure.

The purpose of this study is to determine whether T-wave alternans, as measured through the lead of an implantable defibrillator, is produced by acute ischemia induced by occlusion during percutaneous coronary interventions.

ELIGIBILITY:
Inclusion Criteria:

* patient with CAD undergoing PCI with appropriate Medtronic implantable defibrillator.

Exclusion Criteria:

* non-elective procedure
* non-qualifying defibrillator type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease (CAD) undergoing PCI that also have an appropriate Medtronic implantable defibrillator.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Dizon, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medtronic Defibrillator
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic Defibrillator
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Positive T Wave Studies During a Coronary Intervention
Description: Positive T wave alternans is determined by a proprietary program using ECG recordings during a stress test. The result is reported as positive, negative, or indeterminate.
Time Frame: During the coronary intervention, upto 2 hours
Population: Only collected on subjects that had an intervention
Measure: Number; unit: participants
Arm/Group | Medtronic Defibrillator
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Arm/Group | Medtronic Defibrillator
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No